CLINICAL TRIAL: NCT02941458
Title: Thoracic Tumours Register
Acronym: RTT
Status: Recruiting | Type: Observational
Sponsor: Spanish Lung Cancer Group (Other)
Responsible Party: Sponsor
Other Study IDs: GECP 16/01_RTT
Record Dates: First submitted 2016-10-19; First posted 2016-10-21 (Estimated); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Thoracic Tumors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Non-small cell lung cancer: patients treated for a non small cell lung cancer
- Small cell lung cancer: patients treated for a small cell lung cancer
- Mesotelioma: patients treated for a mesotelioma
- timic cancer: patients treated for a timic cancer
- carcinoid cancer: patients treated for a carcinoid cancer

SUMMARY:
Observational, multicenter study in patients with lung cancer and other thoracic tumors.

The GECP, in its commitment to improve the treatment and prognosis of patients with lung cancer and other thoracic tumors, has marked the individualization of treatment according to the expression of markers predictive of response to chemotherapeutic agents and molecular inhibitors of cell proliferation as one of its primary objectives. This could significantly improve the prognosis of patients with lung cancer, and will lead to a radical change in routine clinical practice. The aim of the register is to explore all data available of all patients treated because of thoracic tumours.

DETAILED DESCRIPTION:
Observational, multicenter study in patients with lung cancer and other thoracic tumors. In a prospective and retrospective way, information will be obtained from the clinical history of each patient.

In Europe, patients with lung cancer have a poor prognosis, and there has been only limited improvement between 1999 and 2007. Potential advantages of the centralization of care and the discussion of treatment strategies in multidisciplinary teams, as suggested in other studies,13 require further research. However, the priorities should be to prevent lung cancer by implementing anti-smoking policies and controlling asbestos exposure throughout Europe, such as was recommended by the World Health Organization (WHO) in 2008.14 Other priorities are to reduce levels of residential radon in risk areas, and early diagnosis to improve the results of surgery, which is still the main curative treatment.

The variability in the diagnostic process, treatment and advocacy, as well as the anticipated increase in associated mortality in Spain in coming years, has stimulated the creation of an epidemiological, observational, multicenter study of cases of lung cancer and other thoracic tumors diagnosed and treated by medical personnel, including both thoracic surgeons and medical oncologists. Data from this study will be collected retrospectively and prospectively, so as to enable an extensive study of the epidemiological and therapeutic factors related to the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thoracic disease, treated with an active treatment or not treated (only palliative care)

Exclusion Criteria:

* Patients with other type of tumours

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients treated due to a thoracic tumour
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-07-21 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Describe epidemiology characteristics of lung cancer and other thoracic tumors in Spanish people | up to 10 years
  To know the epidemiology characteristics of lung cancer and other thoracic tumors in Spain, as well as clinical and histological data, diagnosis, treatments received, and prognostic factors

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Principal Investigator — Hospital Puerta del Hierro
Locations (79):
- Spain (79):
  - Complejo Hospitalario Universitario de Ferrol, Ferrol, A Coruña
  - H. Virgen de los Lirios, Alcoy, Alicante
  - Hospital de Elche, Elche, Alicante
  - Hospital General de Elda, Elda, Alicante
  - H. Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de Granollers, Granollers, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Hospital General La Mancha Centro, Alcázar de San Juan, Ciudad Real
  - Complejo Hospitalario de la Coruña, A Coruña, Coruña
  - H. Insular de Gran Canarias, Las Palmas de Gran Canaria, Gran Canarias
  - Hospital Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital HLA Moncloa, Aravaca, Madrid
  - H. Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario de Móstoles, Móstoles, Madrid
  - Hospital Universitario Infanta Cristina, Parla, Madrid
  - Hospital Universitario Quirón Madrid, Pozuelo de Alarcón, Madrid
  - Hospital General Universitario Santa Lucía, Cartagena, Murcia
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Reina Sofía, Tudela, Navarre
  - Complejo Hospitalario de Vigo, Vigo, Pontevedra
  - Hospital Sant Joan de Reus, Reus, Tarragona
  - Hospital Verge de la Cinta, Tortosa, Tarragona
  - H. Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital Universitari de la Ribera, Alzira, Valencia
  - Hospital Lluís Alcanyís, Xàtiva, Valencia
  - Hospital de Basurto, Bilbao, Vizcaya
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital General de Alicante, Alicante
  - Clinica Tres Torres, Barcelona
  - IOB Hospital Quirón Salud Barcelona, Barcelona
  - HM Hospital Ntra. Sra. de la Esperanza, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital de Burgos, Burgos
  - H. Provincial de Castellón, Castelló
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital Virgen de la Luz, Cuenca
  - H. de Donostia, Donostia / San Sebastian
  - Hospital Dr. Josep Trueta, Girona
  - H. Virgen de las Nieves, Granada
  - Oncogranada, Granada
  - Hospital Universitari de Guadalajara, Guadalajara
  - Hospital de Jaén, Jaén
  - Complejo Asistencial Universitario de León, León
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital La Princesa, Madrid
  - H.U. Puerta de Hierro, Madrid
  - Fundación Jimenez Diaz, Madrid
  - Imoncology, Madrid
  - Hospital Universitario Sanchinarro, Madrid
  - Hospital Universitario Infanta Sofía, Madrid
  - H. Clínico San Carlos, Madrid
  - H. La Paz, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Quirón Salud Málaga, Málaga
  - H. Carlos Haya, Málaga
  - Hospital Virgen de la Victoria, Málaga
  - H. Morales Messeguer, Murcia
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Santa María Naí, Ourense
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Clinico de Salamanca, Salamanca
  - Hospital Nuestra Señora Candelaria, Santa Cruz de Tenerife
  - Hospital de Segovia, Segovia
  - Hospital Virgen del Rocío, Seville
  - Hospital Sant Pau i Santa Tecla, Tarragona
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona
  - Hospital Virgen de la Salud, Toledo
  - Instituto Valenciano de Oncología, Valencia
  - H. General U. de Valencia, Valencia
  - H. Arnau de Vilanova Valencia, Valencia
  - Hospital Dr. Peset, Valencia
  - Hospital La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Complejo Asistencial de Zamora, Zamora
  - Hospital Universitario de Áraba, Vitoria-Gasteiz, Áraba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Provencio M, Cobo M, Rodriguez-Abreu D, Carcereny E, Calvo V, Castro RL, Bernabe R, Bruno MF, Bosch-Barrera J, Barco ED, Medina K, Sanchez-Hernandez A, Suay G, Ortega AL, Vazquez S, Lazaro-Quintela M, Guirado M, Estival A, Blanco M, Cantero A, Massuti B. Biomarker landscape in advanced NSCLC: insights from a national prospective registry. Lung Cancer. 2025 Sep;207:108680. doi: 10.1016/j.lungcan.2025.108680. Epub 2025 Jul 28. PMID 40749260
- [Derived] Provencio M, Cobo M, Rodriguez-Abreu D, Carcereny E, Cantero A, Calvo V, Lopez Castro R, Bernabe R, Bosch-Barrera J, Massuti B, Garcia Campelo R, Sanchez-Hernandez A, Laura Ortega A, Guirado M, Del Barco E, Camps C, Casal-Rubio J, Domine M, Angeles Sala M, Padilla A, Luis Gonzalez Larriba J, de Asis Aparisi F; Spanish Lung Cancer Group SLCG/GECP. Describing differences among populations of thoracic tumors patients under and over 80 years: Data analysis from the SLCG thoracic tumor registry. Lung Cancer. 2024 Apr;190:107513. doi: 10.1016/j.lungcan.2024.107513. Epub 2024 Feb 29. PMID 38432027
- See also: Related Info — http://www.gecp.org